CLINICAL TRIAL: NCT03646955
Title: The DBCG RT Natural Trial: Partial Breast Versus no Irradiation for Women >=60 Years Operated With Breast Conservation for an Early Breast Cancer: a Clinically Controlled Randomized Phase III Trial
Brief Title: Partial Breast Versus no Irradiation for Women With Early Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Collaborators: Danish Cancer Society (Other); Danish Center for Interventional Research in Radiation Oncology (CIRRO) (Other)
Responsible Party: Principal Investigator, Birgitte Offersen, Professor, PhD, MD, Danish Breast Cancer Cooperative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBCG RT Natural Trial
Record Dates: First submitted 2018-07-14; First posted 2018-08-24 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Local Neoplasm Recurrence; Distantly Metastatic Malignant Neoplasm; Death; Fibrosis Breast; Depigmentation/Hyperpigmentation of Skin; Telangiectasia; Scar; Pain; PROMs
MeSH Terms: conditions — Neoplasm Recurrence, Local; Death; Vitiligo; Hyperpigmentation; Telangiectasis; Cicatrix; Pain

STUDY DESIGN:
Intervention Model Description: Clinically controlled randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial breast irradiation (Active Comparator): External beam irradiation 40 Gy / 15 fractions, 5 fractions per week, 3 weeks
  Interventions: Radiation: No partial breast irradiation
- No partial breast irradiation (No Intervention): No radiation therapy

INTERVENTIONS:
Radiation: No partial breast irradiation — Omission of radiation therapy
  Arms: Partial breast irradiation

SUMMARY:
All early breast cancer patients are offered adjuvant breast radiation therapy (RT) after breast conserving surgery for an early breast cancer. Breast cancer is heterogeneous, and selected patients have a very low gain from RT, whilst they still have risk of acute and late side effects from RT. This trial will try identify selection criteria for low risk breast cancer patients who can safely omit adjuvant RT without unacceptable high risk of local failure.

DETAILED DESCRIPTION:
International standard of therapy is to provide adjuvant breast radiation therapy (RT) after breast conserving surgery for an early breast cancer to lower the risk of local and distant failures. However, breast cancer is a heterogeneous disease, and the gain from RT in selected low risk patients is low. RT may cause acute and late side effects, and some of these may be serious to the patient. Therefore, there is a need to tailor RT utilization to the individual recurrence risk and try identify patients who are unlikely to gain much risk reduction from RT, because those patients can then omit RT and thereby avoid late effects and over-treatment. At the present time there is no consensus as to define the selection criteria for patients who may omit RT.

Based on early results from the randomized DBCG RT PBI trial, external beam 40 Gy/15 fr partial breast irradiation (PBI) has been standard in Denmark since April 2016 for selected low risk breast cancer patients. Based on results from the UK IMPORT LOW trial, the 5 yr local recurrence risk using this technique for PBI is 0.5%, whilst 2% for developing a new contralateral breast cancer.

This trial will investigate if PBI can safely be omitted in selected low risk breast cancer patients without causing unacceptable high risk of local failure.

ELIGIBILITY:
Inclusion Criteria:

Female patient >=60 years

Primary tumour characteristics by conventional histopathology

* unilateral and unifocal non-lobular histology grade 1-2
* maximum microscopic size <=20mm
* node negative determined by sentinel node or axillary lymph node dissection
* estrogen receptor >=10% positive
* HER2 negative (by IHC and/or in situ hybridization)
* resection margin >=2 mm for invasive carcinoma and any ductal carcinoma in situ associated with the cancer

Surgical type is breast conservation

Performance status ECOG 0-2

No evidence of distant metastasis

Exclusion Criteria:

* multifocal or multicentric invasive carcinoma or ductal carcinoma in situ
* evidence of clinical or pathological T4 breast cancer
* grade 3 malignancy
* previous breast cancer or DCIS irrespective of disease-free interval
* previous radiation therapy to the breast or thorax,
* previous neoplasm within 5 years except carcinoma in situ of the cervix, endometrium or coli, melanoma in situ.
* comorbidity precluding the patient from radiation therapy (e.g. cardiovascular or pulmonary disease, scleroderma, systemic lupus erythematosus).
* mental/psychiatric disorder which precludes the patient from understanding the randomization and the follow up.
* documented hereditary breast cancer or with high genetic risk of breast cancer
* life expectancy <10 years

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 926 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2033-09-01 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
Invasive local recurrence | 10 years
  Invasive local recurrence

SECONDARY OUTCOMES:
Regional nodes recurrence | 10 years
  Invasive recurrence in regional nodes of the treated breast
Distant failure | 10 years
  Invasive recurrence from the breast cancer outside the loco-regional area
Death | 10 years
  Death and cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte V Offersen, PhD, Principal Investigator — Danish Breast Cancer Group
Locations (17):
- Ponticia Universidad Catolica de Chile, Santiago, Chile
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Naestved Hospital, Næstved
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle
- Norway (6):
  - Haukeland HUS, Bergen
  - Nordlandssykehuset, Bodø
  - Kristiansand Hospital, Kristiansand
  - Oslo University Hospital, Radiumhospitalet, Oslo
  - Stavanger Hospital, Stavanger
  - Tromsø University Hospital, Tromsø
- Sweden (3):
  - Sahlgrenska University hospital, Gothenburg
  - Skånes University Hospital, Lund
  - Uppsala Akademiska Sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
When the results from the trial are published, the DBCG RT Committee can decide that the results may be part of a meta-analysis.
Supporting Information: Study Protocol
Time Frame: It will only be possible if the DBCG Radiation Therapy Committee decides that it is acceptable
Access Criteria: The DBCG Radiation Therapy Committee will define the criteria after publication of the results from the trial